CLINICAL TRIAL: NCT04366479
Title: Effect of Endurance Exercise on nrf2 mRNA Expression Gene and Physical Fitness (VO2max) of Indonesian Hajj Health Officers
Brief Title: Endurance Exercise on nrf2 mRNA Expression Gene and VO2max
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Collaborators: Indonesia-MoH (Other Government)
Responsible Party: Principal Investigator, Ismail Ahmad, Associate Professor, Hasanuddin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HasanuddinU
Record Dates: First submitted 2020-04-17; First posted 2020-04-29 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Physical Fitness
Keywords: Endurance Exercise; Nuclear Respiratory Factor; Physical Fitness (VO2max)

STUDY DESIGN:
Intervention Model Description: This type of quasi-experimental research (quasy experiment) with pre-test and post-test research design with only control design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): The study lasted for 5 weeks (1 month 7 days). During the research process, we monitor closely, especially the training schedule, implementation, and evaluation, directly and indirectly. Directly assisting participants to do endurance training activities, not directly monitoring via telephone or WhatsApp.
  Interventions: Behavioral: Multistage Fitness Test

INTERVENTIONS:
Behavioral: Multistage Fitness Test — Participants only joined in one group will be given intervention for 5 weeks in the form of running 1600 meters duration of 20-30 minutes 3 times a week. It is important for the participants as well as for us to know which training methods are given. this information will be documented in our file, but we will not see these files until after the research is complete. this is the best way we have for testing without being influenced by what we think or expect might happen.

SUMMARY:
Indonesian Hajj Health Officers have the responsibility and very important role in providing health services for Indonesian pilgrims during embarkation and debarkation. One of the main indicators of success is they have excellent physical fitness. This study aims to determine the effectiveness of an intervention program by comparing the results of (intervention) intervention groups, namely the effect of physical exercise interventions (endurance exercise) measured before and after the intervention. This research is an intervention study, and I understand that the process of taking blood can occur with fear, pain due to being pricked by a needle, can faint or be infected. However, previous blood pressure tests, sterile collection techniques and performed by experts, are very unlikely to cause side effects.

DETAILED DESCRIPTION:
The investigators invite all Indonesian Hajj Health Officers candidates to participate in research on physical fitness (VO2max) which is an important part of providing Hajj health services in Saudi Arabia while they are on duty. I was involved in the RT-PCR examination and physical fitness test (VO2max) that was carried out before the intervention program and was briefed on the examination protocol before being tested. The consent form was given to me first to be handled. I was informed about the intervention process and the purpose of the research, as well as the confidentiality of the data, collected. And it was also stated that I would be allowed to withdraw from the research at any time without pressure and coercion from any party. The procedure investigators will do is take samples from prospective Indonesian Hajj Health Officers undergoing a series of anamneses and physical examinations by doctors, in the form of personal data, physical activities, general physical examinations including TB, BB, HR, RR, then performed the physical activity eligibility forms. Next, a 1 ml blood sample is taken into a purple test tube containing EDTA to prevent lysis. The blood sample is taken to the HUM-RC Makassar Biomolecular Biology laboratory and stored in a frozen cupboard, after which an initial physical fitness measurement (VO2max) test is carried out using the Multi Fitness Test (MFT) or Bleep Test to PRE TEST at the Health Training Center (Health Training Center) BBPK) Makassar, followed by running exercises intervention as far as 1600 meters 3 times a week duration of 20-30 each training session with a frequency of exercise 16 times 5 weeks according to a predetermined schedule, then conducted a physical fitness test (VO2max) using the same method when PRE TEST to POST TEST I, followed by 1 ml blood sampling at Sudiang Embarkation Hajj Makassar, then 1 week later physical fitness test (VO2max) to POST TEST II without blood sampling is taken again.

Participants (n = 30), measured physical fitness level (VO2max) using the Multistage Fitness Test (MFT) Bleep Test (level and feedback) method before being given intervention (pre-exercise), after that given a running intervention 1600 meters duration 20 -30 minutes each training session 3 times a week with a frequency of exercise16 times for 5 weeks, then physical fitness measurements (VO2max) → (post-exercise 1), then intermittent 1-week duration of physical fitness measurements (VO2max) again without intervention and blood sampling (post-exercise 2).

Participants only joined in one group will be given intervention for 5 weeks in the form of running 1600 meters duration of 20-30 minutes 3 times a week. It is important for the participants as well as for us to know which training methods are given. this information will be documented in our file, but the investigators will not see these files until after the research is complete. this is the best way the investigators have for testing without being influenced by what the investigators think or expect might happen.

The doctor in charge of research will always look after the participants very carefully during the study. If the investigators are worried about what is done, the investigators will find out how the level of physical fitness that participants get and make changes. If there is something the participant is worried about or is disturbing the Participant about the research, please talk to me or one of the other researchers.

In this study, the investigators did not use a placebo term, but the investigators still explained to participants in the world of research that the term placebo is known as clinical trials or interventions given to participants that are not genuine but fake. For good research, participants mustn't know whether the participants have been properly measured according to the criteria or not. This is one of the best ways the investigators have to find out what level of physical fitness the investigators are testing. No side effects might occur because the previous sample was very rigorously selected through analysis, physical examination and physical activity feasibility testing. If Participants find that Our interventions are very uncomfortable for participants, the investigators can use other exercise options more comfortably according to the available exercise choices.

The possibility of danger, risk, or side effects in this study is very small because the selection of samples is done very closely starting with anamnesis and head-to-toe physical examination and continued with a physical activity feasibility test (PAR-Q). If the physical fitness test occurs when there is suffocation, the researcher has prepared 2 medical staff who accompanied the subjects during the physical fitness test and also in this study the investigators prepared 2 clinics namely the Makassar BBPK Health Clinic which was used during the physical fitness pre-test and the Clinic Musytasyfa Health Makassar Haji Sudiang Dormitory that was used at the time of physical fitness post-test.

During the study, the investigators carried out a series of research processes as follows: Pre-exercise

* In the first stage: Conducting anamneses and physical examinations by doctors, in the form of personal data, physical activity, general physical examination including Height, Weight, Heart Rate, Respiratory Rate, Blood Pressure (BP)
* In the second stage: Completion of physical activity eligibility forms.
* In the third step: a 1 ml blood sample is taken into a purple test tube containing EDTA to prevent lysis. The blood samples were taken to the Makassar HUM-RC Biomolecular Biology laboratory and stored in a frozen cupboard.
* In the fourth step: Measurement of the initial physical fitness test (VO2max) using the Multi Fitness Test (MFT) or Bleep Test to PRE TEST at the Makassar Health Training Center (BBPK) Endurance Exercise
* In the first stage: Selecting an exercise schedule according to the provisions of the study
* In the second stage: Exercise choice I: Monday-Wednesday-Friday; Exercise choice II: Tuesday-Thursday-Saturday; Exercise choice III: Wednesday-Friday-Sunday
* In the third stage: Document endurance exercises in the form of a video exercise Post Exercise I
* In the first stage: Initial physical fitness test (VO2max) measurement using the Multi Fitness Test (MFT) or Bleep Test to POST TEST I at the Haji Sudiang Makassar Dormitory In the second stage: Recovery 1 hour after the physical fitness test In the third stage: Taking 1 ml of blood sample inserted in a purple test tube containing EDTA to prevent lysis. The blood samples were taken to the Makassar HUM-RC Biomolecular Biology laboratory and stored in a frozen cupboard.

Post Exercise II Measurement of the initial physical fitness test (VO2max) using the Multi Fitness Test (MFT) or Bleep Test to POST TEST II at the Makassar Sports Hall

ELIGIBILITY:
Inclusion Criteria:

* Participants from the Nurse profession aged 30 - 39 years
* Pass the selection of candidates for Indonesian Hajj Health Officers
* Understand the physical training program instructions in the rockport method
* Willing to participate in activities and all research provisions

Exclusion Criteria:

* Had a history of coronary heart disease,asthma
* Not approved by the doctor to participate in the study due to a medical condition

Ages: 30 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
VO2max Measurement | 5 weeks
  Aerobic capacity is also known as maximal oxygen uptake or maximum oxygen consumption (VO2max)
Measurement of mRNA NRF2 Gene Expression | 5 weeks
  RT-PCR analyzes human RNA in the nrf2 RNA sample as the target gene and GAPDH is selected as the housekeeping gene

CONTACTS AND LOCATIONS:
Overall Officials: Mochammad Hatta, Profesor, Principal Investigator — Department of Biomolecular Medicine, Hasanuddin University Makassar
Locations (1):
- Makassar Center for Health Training, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vivian H. Heyward. (2016). Aerobic Capacity, Physical Fitness and VO2 Maxium Measurement. Advance Fitness Assessment & Exercise Prescription, 252(805), 2-5. https://www.biopac.com/wp-content/uploads/app252.pdf
- [Result] Lockie RG, Dawes JJ, Moreno MR, Cesario KA, Balfany K, Stierli M, Dulla JM, Orr RM. Relationship Between the 20-m Multistage Fitness Test and 2.4-km Run in Law Enforcement Recruits. J Strength Cond Res. 2021 Oct 1;35(10):2756-2761. doi: 10.1519/JSC.0000000000003217. PMID 31268997
- [Result] Zhao XQ, Zhang YF, Xia YF, Zhou ZM, Cao YQ. Promoter demethylation of nuclear factor-erythroid 2-related factor 2 gene in drug-resistant colon cancer cells. Oncol Lett. 2015 Sep;10(3):1287-1292. doi: 10.3892/ol.2015.3468. Epub 2015 Jul 8. PMID 26622665

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT04366479/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT04366479/ICF_001.pdf